CLINICAL TRIAL: NCT02965391
Title: Dynamic Changes and Surveillance of Circulating Tumor DNA in Surgical Non-small Cell Lung Cancer Patients
Brief Title: Dynamic Changes of Circulating Tumor DNA in Surgical Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Chen KeZhong, Principal Investigator, Peking University People's Hospital
Other Study IDs: PTHO1602
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma; Non-small-cell Lung Cancer; Lung Neoplasms
Keywords: Circulating Tumor DNA; Half time; Lung cancer; Surgery; Surveillance
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — A series of lung cancer patients plasma before or after surgery.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Previous study showed circulating tumor DNA levels reflect the total systemic tumor burden. Circulating tumor DNA levels should decrease after complete surgery and could be increase as tumor recurrence. Few study investigated the half time of circulating tumor DNA in lung cancer patients that no criterion has been established of how to use it for surveillance.

DETAILED DESCRIPTION:
For lung cancer patients who received surgery, multiple time of plasma will be collected before or after surgery. A series of mutations will be detected in plasma before surgery based on next generation sequencing. The positive mutation will be traced after surgery and in follow up.

ELIGIBILITY:
Inclusion Criteria:

* Suspected lung cancer before surgery
* No malignant tumor history within the past 5 years
* The pulmonary nodule is not pure ground glass opacity
* Patients must have given written informed consent

Exclusion Criteria:

* Multiple primary lung cancer
* R1,R2 resection
* Histology confirmed not non-small cell lung cancer
* Unqualified blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed lung cancer patients who received completely tumor resection
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Half-life of circulating tumor DNA after surgery | 3 months

SECONDARY OUTCOMES:
The variation of circulating tumor DNA level before and after surgery | 3 months
Correlation of circulating tumor DNA level after surgery with tumor recurrence | 3 years
Correlation of circulating tumor DNA level after surgery with clinical features | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, M.D., Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen K, Zhao H, Shi Y, Yang F, Wang LT, Kang G, Nie Y, Wang J. Perioperative Dynamic Changes in Circulating Tumor DNA in Patients with Lung Cancer (DYNAMIC). Clin Cancer Res. 2019 Dec 1;25(23):7058-7067. doi: 10.1158/1078-0432.CCR-19-1213. Epub 2019 Aug 22. PMID 31439586
- [Derived] Chen K, Zhao H, Yang F, Hui B, Wang T, Wang LT, Shi Y, Wang J. Dynamic changes of circulating tumour DNA in surgical lung cancer patients: protocol for a prospective observational study. BMJ Open. 2018 Feb 6;8(2):e019012. doi: 10.1136/bmjopen-2017-019012. PMID 29437753